CLINICAL TRIAL: NCT03159507
Title: Effect of Omega-3 Index on Cellular Metabolism and Quality of Life Following the Administration of a Customized Dose of Omega-3 Oil
Brief Title: Effect of Omega-3 Index on Cellular Metabolism and Quality of Life
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SCF Pharma (Industry)
Collaborators: Université du Québec à Rimouski (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IO3-01
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Omega-3 Index; Cellular metabolism; EPA Monoglyceride; Quality of life
MeSH Terms: interventions — 1-eicosapentaenoylglycerol

STUDY DESIGN:
Intervention Model Description: Prospective, single arm trial where each participant receives a personalized dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAG-EPA (Experimental): MAG-EPA softgel (500mg), daily dose between 1g and 3.5g
  Interventions: Dietary Supplement: MAG-EPA

INTERVENTIONS:
Dietary Supplement: MAG-EPA — Based on the result of the participant's Omega-3 index obtained from the blood sampling of visit 1, the daily dose of MAG-EPA will be adjusted to obtain an Omega-3 Index of 8.

SUMMARY:
Determine whether personal optimization of the Omega-3 index improves cellular metabolism and quality of life (according to the SF-36 form).

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 19 or over
* Available for the entire duration of the study and willing to participate on the basis of the information provided in the FIU duly read and signed.

Exclusion Criteria:

* Allergy known to fish
* Pregnant women who breast-feed or test positive for pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Omega-3 Index | 8 weeks
  Achievement of an omega-3 index of 8.

SECONDARY OUTCOMES:
Cellular metabolism | 8 weeks
  To determine whether the achievement of the optimal level of the omega-3 index results in an improvement in the white blood cell energy metabolism
Quality of life | 8 weeks
  Determine whether the achievement of the optimal level of the Omega-3 index results in an improvement in quality of life (according to Form SF-36)
Heart rate | 8 weeks
  Confirm the link between the optimal omega-3 index and heart rate (bpm)
Total Cholesterol | 8 weeks
  Confirm the link between the optimal omega-3 index and total cholesterol (in mmol/L)
Triglycerides | 8 weeks
  Confirm the link between the optimal omega-3 index and triglycerides level (in mmol/L)
HDL-cholesterol | 8 weeks
  Confirm the link between the optimal omega-3 index and HDL-cholesterol (in mmol/L)
LDL-cholesterol | 8 weeks
  Confirm the link between the optimal omega-3 index and LDL-cholesterol (in mmol/L)
Alanine aminotransferase | 8 weeks
  Confirm the link between the optimal omega-3 index and alanine aminotransferase (in U/L
Aspartate aminotransferase | 8 weeks
  Confirm the link between the optimal omega-3 index and aspartate aminotransferase (in U/L)
Bilirubin | 8 weeks
  Confirm the link between the optimal omega-3 index and Bilirubin (in µmol/L)
Albumin | 8 weeks
  Confirm the link between the optimal omega-3 index and Albumin (in g/L)
C-reactive protein | 8 weeks
  Confirm the link between the optimal omega-3 index and C-reactive protein (in mg/L)
Apolipoprotein B | 8 weeks
  Confirm the link between the optimal omega-3 index and Apolipoprotin B (in mmol/L)
Erythrocyte sedimentation rate | 8 weeks
  Confirm the link between the optimal omega-3 index and the erythrocyte sedimentation rate (in min)
Systolic blood pressure | 8 weeks
  Confirm the link between the optimal omega-3 index and the systolic blood pressure (in mm Hg)
Diastolic blood pressure | 8 weeks
  Confirm the link between the optimal omega-3 index and the diastolic blood pressure (in mm Hg)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Julie Landry, MSc, Study Director — SCF Pharma
Locations (1):
- SCF Pharma, Rimouski, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No